CLINICAL TRIAL: NCT03615365
Title: Characterisation of COPD Breathing Records During Exacerbations
Brief Title: COPD Breathing Record Study 2
Acronym: CBRS2
Status: Completed | Type: Observational
Sponsor: TidalSense (Industry)
Responsible Party: Sponsor
Other Study IDs: G007-17_CBRS2
Record Dates: First submitted 2018-07-19; First posted 2018-08-03 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2018-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Capnography; Diagnosis; Breathlessness; Exacerbations; Device
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Disease; Dyspnea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with moderate-to-severe COPD.: Patients will be identified from the Cambridge COPD Centre. This unit sees patients following emergency admissions, GP referrals and has a regional referral base for complex COPD. Patients' medical records will be reviewed and classified according to GOLD criteria.
  Patients will undergo a clinical assessment of COPD during screening at Addenbrooke's Hospital. All patients will be assessed five times: at the start, 2 weeks, 10 weeks, 18 weeks and at the end of the 26 week study period. A brief follow-up telephone review will be conducted approximately 2 weeks after the end of the monitoring period. At each assessment, capnometry measurements will be taken in addition to vital signs and pulse oximetry.

SUMMARY:
The aim of this study is to collect capnometric (tidal breathing CO2) data using TidalSense's N-Tidal C Data Collector Device. The data collected will be examined for correlation with currently accepted assessment techniques for COPD (spirometry, vital signs and pulse oximetry) and the patient's clinical condition (stable, worsening, improving). The patient numbers and study duration have been determined by power calculations to provide a statistically significant sample size, based on expected number of exacerbations (mild, moderate and severe) from the patient cohort. The data will also be examined to assess the predictive possibility of a non-invasive self-care personal CO2 monitoring device to identify COPD exacerbations.

DETAILED DESCRIPTION:
Study Design: This is an uncontrolled, non-randomised, un-blinded longitudinal observational data collection study with the N-Tidal C Data Collector Device in patients with COPD.

Patients will be identified from the Cambridge COPD Centre. This unit sees patients following emergency admissions, GP referrals and has a regional referral base for complex COPD. Patients' medical records will be reviewed and classified according to GOLD criteria. Those patients who are classified as COPD with appropriate inclusion criteria (below) will be invited to participate. Patients who give informed consent will be screened for the study.

The N-Tidal C Data Collector Device will be explained to the patients and they will be trained how to use it. All patients will complete a short daily diary record.

Patients will undergo a clinical assessment of COPD during screening at Addenbrooke's Hospital. All patients will be assessed five times: at the start, 2 weeks, 10 weeks, 18 weeks and at the end of the 26 week study period. A brief follow-up telephone review will be conducted approximately 2 weeks after the end of the monitoring period. At each assessment, capnometry measurements will be taken in addition to vital signs and pulse oximetry. The study will not interfere with routine management of the patient's condition.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 40 years and over.
2. Diagnosis of COPD (Primary) and at least one moderate exacerbation within 12 months of the start of the study period.
3. Able to provide signed informed consent.

Exclusion Criteria:

1. Patients who, in the opinion of the investigator, are unlikely to comply with the requirements of the study, use the device correctly or keep the diary records;
2. Diagnosis of neuromuscular disorders or Kyphoscoliosis;
3. Diagnosis of other Respiratory disorders that, in the opinion of the investigator, would impact the conduct of the study e.g. clinically significant bronchiectasis, asthma;
4. Patients who have experienced an exacerbation of their COPD that has required treatment with antibiotics and/or oral corticosteroids within 2 weeks prior to the study start.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate-to-severe chronic obstructive pulmonary disease (COPD) will be identified from the Cambridge COPD Centre.
  Those patients with COPD satisfying the inclusion criteria will be invited to participate.
  The majority of these will be GOLD D.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2018-11-23 (Actual)

PRIMARY OUTCOMES:
To measure the changes in the α angle of the tidal breathing CO2 (TBCO2) waveform data from stable COPD through an exacerbation and back to stable. | Throughout the 26 week use of the N-Tidal C device for each patient.
  The α angle is one of the key parameters extracted from the TBCO2 waveform data captured by the N-Tidal C device.
  The α angle is given in degrees and significant changes in the α angle have previously been observed between stable COPD and acute exacerbations of COPD.
To measure the minimum and maximum CO2 levels of the TBCO2 waveform data from stable COPD through an exacerbation and back to stable. | Throughout the 26 week use of the N-Tidal C device for each patient.
  The minimum and maximum CO2 levels are key parameters extracted from the TBCO2 waveform data captured by the N-Tidal C device.
  CO2 levels are given in kPa and significant differences have previously been observed between stable COPD and acute exacerbations of COPD.
To measure the variability of breath length of the TBCO2 waveform data from stable COPD through an exacerbation and back to stable. | Throughout the 26 week use of the N-Tidal C device for each patient.
  The variability of breath length is one of the key parameters extracted from the TBCO2 waveform data captured by the N-Tidal C device.
  Breath length is measured in seconds and significant differences have previously been observed between stable COPD and acute exacerbations of COPD.
To measure the standard deviation of End Tidal CO2 levels of the TBCO2 waveform data from stable COPD through an exacerbation and back to stable. | Throughout the 26 week use of the N-Tidal C device for each patient.
  The standard deviation of End Tidal CO2 levels is one of the key parameters extracted from the TBCO2 waveform data captured by the N-Tidal C device.
  End Tidal CO2 levels are given in kPa and significant differences have previously been observed between stable COPD and acute exacerbations of COPD.

SECONDARY OUTCOMES:
Longitudinal Database | Throughout the 26 week use of the N-Tidal C device for each patient.
  To collect a longitudinal observational database of TBCO2 waveform records for up to 50 patients with COPD over a period of 26 weeks using the N-Tidal C device.
COPD Exacerbations | Throughout the 26 week use of the N-Tidal C device for each patient.
  To capture the carbon dioxide signature predictive of exacerbations in monitored patients who undergo mild, moderate and severe exacerbations during the study.
COPD Variability | Throughout the 26 week use of the N-Tidal C device for each patient.
  To identify the within-day and day-to-day variability of respired CO2 in patients with COPD
Usability of the N-Tidal C device | Throughout the 26 week use of the N-Tidal C device for each patient.
  Measured by the patients compliance and perseverance to the use the N-Tidal C device.
Acceptability of the N-Tidal C device | At the end of the 26 week use of the N-Tidal C device for each patient.
  The patients will be asked questions about the ease of use of the N-Tidal C and twice daily respiratory monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Mahadeva, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Addenbrooke's Hospital, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Talker L, Neville D, Wiffen L, Selim AB, Haines M, Carter JC, Broomfield H, Lim RH, Lambert G; BRS Study Team; Weiss ST, Hayward G, Brown T, Chauhan A, Patel AX. Machine diagnosis of chronic obstructive pulmonary disease using a novel fast-response capnometer. Respir Res. 2023 Jun 2;24(1):150. doi: 10.1186/s12931-023-02460-z. PMID 37268935